CLINICAL TRIAL: NCT04313127
Title: A Single-center,Open-label，Dose-escalating Phase I Clinical Trial to Evaluate Recombinant Novel Coronavirus Vaccine (Adenovirus Type 5 Vector) in Healthy Adults Aged 18-60 Years Old
Brief Title: Phase I Clinical Trial of a COVID-19 Vaccine in 18-60 Healthy Adults
Acronym: CTCOVID-19
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CanSino Biologics Inc. (Industry)
Collaborators: Institute of Biotechnology, Academy of Military Medical Sciences, PLA of China (Other); Jiangsu Province Centers for Disease Control and Prevention (Network); Hubei Provincial Center for Disease Control and Prevention (Other); Tongji Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: JSVCT088
Record Dates: First submitted 2020-03-15; First posted 2020-03-18 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2020-05

CONDITIONS: COVID-19
Keywords: COVID-19; vaccine; Ad5; Safety; Immunogenicity; Infection; novel coronavirus; Dose-escalation
MeSH Terms: conditions — COVID-19; Alzheimer Disease 5; Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low-dose Group (Experimental): Subjects received one dose of 5E10 vp Ad5-nCoV at 18 to 60 years old
  Interventions: Biological: Recombinant Novel Coronavirus Vaccine (Adenovirus Type 5 Vector)
- Middle-dose Group (Experimental): Subjects received one dose of 1E11 vp Ad5-nCoV at 18 to 60 years old
  Interventions: Biological: Recombinant Novel Coronavirus Vaccine (Adenovirus Type 5 Vector)
- High-dose Group (Experimental): Subjects received one dose of 1.5E11vp Ad5-nCoV at 18 to 60 years old
  Interventions: Biological: Recombinant Novel Coronavirus Vaccine (Adenovirus Type 5 Vector)

INTERVENTIONS:
Biological: Recombinant Novel Coronavirus Vaccine (Adenovirus Type 5 Vector) — Intramuscular other name:Ad5-nCoV

SUMMARY:
The 2019 novel-coronavirus (2019-nCov) is the cause of a cluster of unexplained pneumonia that started in Hubei province in China. It has manifest into a global health crisis with escalating confirmed cases and spread across many countries.

In view of the fact that there is currently no effective antiviral therapy, the prevention or treatment of diseases caused by COVID-19 can be tough for current treatment.

This study is a phase I clinical trial. The investigators intent to evaluate the safety, reactogenicity and immunogenicity of Recombinant Novel Coronavirus Vaccine (Adenovirus Type 5 Vector) .

DETAILED DESCRIPTION:
This is a single-center,open-label，dose-escalating phase I clinical trial in healthy 18 to 60 years of age, inclusive, who are in good health and meet all eligibility criteria. This clinical trial is designed to assess the safety, reactogenicity and immunogenicity of Recombinant Novel Coronavirus Vaccine (Adenovirus Type 5 Vector) manufactured by Beijing Institute of Biotechnology and CanSino Biologics Inc.One hundred and eight subjects will be enrolled into one of three cohorts and will receive an intramuscular (IM) injection of experimental vaccine or placebo on Days 1 in the deltoid muscle.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 60 years.
* Able to understand the content of informed consent and willing to sign the informed consent
* Able and willing to complete all the secluded study process during the whole 6 months study follow-up period.
* Negative in HIV diagnostic test.
* Negative in serum antibodies (IgG and IgM) screening of COVID-19.
* Normal in lung CT images (no imaging features of COVID-19
* Axillary temperature ≤37.0°C.
* The BMI index is 18.5-30.0.
* Negative in Nasopharyngeal swabs / sputum and anal swabs through RT-PCR
* Laboratory tests such as hematological examination and clinical biochemistry examination are in the normal range or without meaning judged by clinical doctor.
* General good health as established by medical history and physical examination.

Exclusion Criteria:

* Family history of seizure, epilepsy, brain or mental disease
* Subject allergic to any component of the investigational vaccine, or a more severe allergic reaction and history of allergies in the past.
* Woman who is pregnant, breast-feeding or positive in β-HCG (human chorionic gonadotropin) pregnancy test (urine) on day of enrollment, or become pregnant during the next 6 months
* Any acute fever disease or infections.
* History of SARS
* Major congenital defects or not well-controlled chronic illness, such as asthma, diabetes, or thyroid disease.
* Serious cardiovascular diseases, such as arrhythmia, conduction block, myocardial infarction, severe hypertension without controllable drugs, etc.
* Hereditary angioneurotic edema or acquired angioneurotic edema
* Urticaria in last one year
* No spleen or functional spleen.
* Platelet disorder or other bleeding disorder may cause injection contraindication
* Faint at the sight of needles.
* Prior administration of immunodepressant or corticosteroids, antianaphylaxis treatment, cytotoxic treatment in last 6 months.
* Prior administration of blood products in last 4 months
* Prior administration of other research medicines in last 1 month
* Prior administration of attenuated vaccine in last 1 month
* Prior administration of inactivated vaccine in last 14 days
* Current anti-tuberculosis prophylaxis or therapy
* According to the judgement of investigator,various medical, psychological, social or other conditions, those could affect the subjects to sign informed consent.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 108 (Actual)
Dates: Start 2020-03-16 (Actual); Primary Completion 2021-01-20 (Actual); Study Completion 2021-02-20 (Actual)

PRIMARY OUTCOMES:
Safety indexes of adverse reactions | 0-7 days post-vaccination
  Occurrence of adverse reactions post-vaccination

SECONDARY OUTCOMES:
Safety indexes of adverse events | 0-28 days post-vaccination
  Occurrence of adverse events post-vaccination
Safety indexes of SAE | 0-28 days, within 6 mouths post-vaccination
  Occurrence of serious adverse events post-vaccination
Safety indexes of lab measures | pre-vaccination, day 7 post-vaccination
  Occurrence of abnormal changes of laboratory safety examinations
Immunogencity indexes of GMT(ELISA) | day14,28，month 3,6 post-vaccination
  Geometric mean titer（GMT）of S-specific antibodies against 2019 novel coronavirus tested by ELISA in serum
Immunogencity indexes of GMT(pseudoviral neutralization test method) | day14,28，month 6 post-vaccination
  Geometric mean titer（GMT）of S-specific antibodies against 2019 novel coronavirus tested by pseudoviral neutralization test method in serum
Immunogencity indexes of seropositivity rates(ELISA) | day14,28，month 3,6 post-vaccination
  the seropositivity rates of S-specific antibodies against 2019 novel coronavirus tested by ELISA in serum
Immunogencity indexes of seropositivity rates(pseudoviral neutralization test method) | day14,28，month 6 post-vaccination
  the seropositivity rates of S-specific antibodies against 2019 novel coronavirus tested by pseudoviral neutralization test method in serum
Immunogencity indexes of GMI(ELISA) | day14,28，month 3,6 post-vaccination
  Geometric mean fold increase（GMI）of S-specific antibodies against 2019 novel coronavirus tested by ELISA in serum
Immunogencity indexes of GMI(pseudoviral neutralization test method) | day14,28，month 6 post-vaccination
  Geometric mean fold increase（GMI）of S-specific antibodies against 2019 novel coronavirus tested by pseudoviral neutralization test method in serum
Immunogencity indexes of GMC(Ad5 vector) | day、14,28，month3,6 post-vaccination
  Geometric mean concentration（GMC）of anti-Ad5 vector neutralizing antibody responses
Immunogencity indexes of GMI(Ad5 vector) | day、14,28，month3,6 post-vaccination
  Geometric mean fold increase（GMI）of anti-Ad5 vector neutralizing antibody responses
Immunogencity indexes of cellular immune | day 14, 28,month 6 post-vaccination
  specific cellular immune responses

OTHER OUTCOMES:
Consistency analysis(ELISA and pseudoviral neutralization test method) | day,14,28, month 6 post-vaccination
  Consistency analysis of S-specific antibodies against 2019 novel coronavirus tested by ELISA against those tested by pseudoviral neutralization test method
Dose-response relationship（Humoral immunity） | day14,28，month 3,6 post-vaccination
  Relationship between Geometric mean titer (GMT) of S protein-specific antibodies against 2019 novel coronavirus and vaccine dose among study groups
Persistence analysis of anti-S protein antibodies | day14,28，month 3,6 post-vaccination
  Persistence analysis of anti-S protein antibodies among study groups
Time-dose-response relationship（Humoral immunity） | day14,28，month 3,6 post-vaccination
  Relationship between the appearance time of S-specific antibodies against 2019 novel coronavirus and the vaccination dose.
Dose-response relationship（ cellular immunity） | day 14, 28,month 6 post-vaccination
  Relationship between cellular immune levels against 2019 novel coronavirus and vaccine dose among study groups
Persistence analysis of cellular immuse | day 14, 28,month 6 post-vaccination
  Persistence analysis of specific cellular immune response
Time-dose-response relationship（cellular immunity） | day 14, 28,month 6 post-vaccination
  Relationship between the appearance time of cellular immunity against 2019 novel coronavirus and the vaccination dose.

CONTACTS AND LOCATIONS:
Overall Officials: Zhu Fengcai, Principal Investigator — Jiangsu Province Centers for Disease Control and Prevention; Guan Xuhua, Principal Investigator — Hubei Provincial Center for Disease Control and Prevention; Wang Wei, Principal Investigator — Tongji Hospital
Locations (1):
- Hubei Provincial Center for Disease Control and Prevention, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Yes
We support data sharing of the individual participant data. The individual participant data that underlie the results reported in this article, after deidentiﬁcation (text, tables, figures, and appendixes) will be shared. Individual participant data will be available beginning 3 months and ending one year following article publication. Supporting clinical documents including study protocol, statistical analysis plan (SAP), and the informed consent form (ICF) will be available immediately following publication for at least one year. Supporting clinical documents access information will be available at http://www.jshealth.com/. Researchers who provide a scientifically sound proposal will be allowed to access to the individual participant data. Proposals should be directed to jszfc@vip.sina.com or cw0226@foxmail.com.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available beginning 3 months and ending one year following article publication
Access Criteria: Data access requests will be reviewed by the sponsor，investigator and collaborators on the basis of scientific merit. To gain access, data requestors will need to sign a data access agreement.
URL: http://www.jshealth.com/

REFERENCES:
- [Derived] Zhu FC, Li YH, Guan XH, Hou LH, Wang WJ, Li JX, Wu SP, Wang BS, Wang Z, Wang L, Jia SY, Jiang HD, Wang L, Jiang T, Hu Y, Gou JB, Xu SB, Xu JJ, Wang XW, Wang W, Chen W. Safety, tolerability, and immunogenicity of a recombinant adenovirus type-5 vectored COVID-19 vaccine: a dose-escalation, open-label, non-randomised, first-in-human trial. Lancet. 2020 Jun 13;395(10240):1845-1854. doi: 10.1016/S0140-6736(20)31208-3. Epub 2020 May 22. PMID 32450106